CLINICAL TRIAL: NCT03317093
Title: Open and Exploratory Trial to Investigate the Pharmacokinetic of Ceftobiprole Medocaril in Patients With CSF Device
Acronym: BASILE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHAVANET BASILEA 2016
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2019-12

CONDITIONS: Inflamed Meninges; Suspected Meningitis; Ventriculitis
MeSH Terms: interventions — ceftobiprole medocaril; Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ceftobiprole Medocaril — 1 single intravenous dose of 500 mg of Mabelio (Ceftobiprole Medocaril) perfused for 2 hours at D0
Other: Blood samples and cerebrospinal fluid — Before and immediately before the end of the perfusion and then at 0.5h, 1h, 3h, 6h, 12h and 24h.

SUMMARY:
Ceftobiprole is a very active new cephalosporin on staphylococci resistant to methicillin (SEMR: Staphylococcus epidermidis Resistant to Meticillin, SAMR: Staphylococcus aureus Resistant to Meticillin) and / or vancomycin; it is also very active on pneumococci resistant to penicillin and / or 3rd generation cephalosporins. This new drug has AMM in nosocomial respiratory infections, Animal work shows the efficacy of ceftobiprole in gram negative bacillus meningeal infections.

The rationale of this study is based on the antibacterial spectrum of ceftobiprole, which would therefore be useful in the treatment of staphylococcal bacterial meningitis resistant patients (SEMR or SAMR) encountered in intensive care and / or neurosurgery and in the treatment of pneumococcal meningitis.

To validate these possibilities, it is necessary to know the concentrations of ceftobiprole in the meningeal space.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years)

  * Provision of informed consent prior to any study specific procedures
  * Female patients of childbearing potential may be entered if pregnancy testing is negative and the patient agrees to abstain from procreational sexual intercourse or must use double-barrier contraceptive measures for the duration of the study
* Presence of an indwelling external CSF access device (ventriculostomy or lumbar drain)
* Presence of inflamed meninges as a result of documented or suspected meningitis or ventriculitis. Patients with both clinical symptoms (fever, headache, meningismus, and altered mentation) and laboratory parameters (CSF leukocytosis, defined as a CSF white blood cell count [WBC] of >103, elevated CSF protein, defined as CSF protein of >1g/l, reduced CSF glucose, defined as CSF glucose of <0.3g/l, or a positive CSF Gram stain or culture) indicative of CNS infection were deemed to have definitive bacterial meningitis/ventriculitis. Inflamed meninges were defined as the presence of >5 leukocytes/mm3 of CSF.
* Person with antibacterial treatment (including treatment for the current meningitis or ventriculitis)
* Glycemia above 3 mmol/l and below 10 mmol/l
* Natremia below 145 mmol/l
* Capnia below 45 mmHg
* No other patient included within 72 hours from D0 (treatment period) of the previous patient
* Agreement of the scientific committee

Exclusion Criteria:

* Hypersensitivity to MABELIO® (ceftobiprole) or to one of its excipient or another 3rd cephalosporin
* Hypersensitivity to cephalosporin
* Immediate and severe hypersensitivity to β-lactam antimicrobial other than Mabelio and other cephalosporins
* Pregnant or breast feeding women
* Renal insufficiency defined as creatinine clearance < 50 mL/min
* Patient with creatinine clearance > 150 mL/min
* Patients with conditions known or suspected to alter pharmacokinetics (i.e., burn or cystic fibrosis patients)
* Refusal to participate
* Person not affiliated to the social security
* Absolute necessity of immediate removing the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Measurement of concentration of ceftobiprole in blood | Before and immediately the end of the perfusion and then at 0.5, 1, 3, 6, 12 and 24 hours
Measurement of concentration of ceftobiprole in cerebrospinal fluid | Before and immediately the end of the perfusion and then at 0.5, 1, 3, 6, 12 and 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France